CLINICAL TRIAL: NCT01302743
Title: Cinnamon Bark, Water-Soluble Cinnamon Extract, and Metformin as Initial Treatment for Type 2 Diabetes Mellitus: A Randomized, Controlled Trial.
Brief Title: Cinnamon Bark, Water-Soluble Cinnamon Extract, and Metformin for Treatment of Type 2 DM.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20110004H
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Diabetes
Keywords: Diabetes; Metformin; Cinnamon
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin (Active Comparator): oral extended-release Metformin 1000 mg once a day for 90 days
  Interventions: Drug: Group 1: Metformin
- Cinnamon Bark (Experimental): Cinnamon Bark 1000 mg once a day for 90 days
  Interventions: Dietary Supplement: Group 2: Cinnamon Bark
- Cinnulin PF (Experimental): Cinnulin PF 500 mg once a day for 90 days
  Interventions: Dietary Supplement: Group 3: Cinnulin PF

INTERVENTIONS:
Drug: Group 1: Metformin — Group 1: Will receive oral extended-release Metformin 1000 mg once a day for 90 days
  Arms: Metformin
Dietary Supplement: Group 2: Cinnamon Bark — Group 2: Will receive Cinnamon Bark 1000 mg once a day for 90 days
  Arms: Cinnamon Bark
Dietary Supplement: Group 3: Cinnulin PF — Group 3: Will receive Cinnulin PF 500 mg once a day for 90 days.
  Arms: Cinnulin PF

SUMMARY:
The purpose of this study is to assess whether Cinnamon bark or water-soluble cinnamon is an effective nutraceutical for the initial treatment of diabetes when compared to standard therapy of Metformin.

DETAILED DESCRIPTION:
We are studying whether or not cinnamon bark or water-soluble cinnamon could be an effective nutraceutical for the initial treatment of diabetes when compared to standard therapy of metformin 1000 mg (extended-release). This study will enroll 309 subjects type 2 diabetics (using American Diabetes Association criteria) on no hypoglycemic medications. Subjects will be randomized into one of three groups, group 1 will receive oral extended-release Metformin 1000mg, group 2 will receive Cinnamon Bark 1000mg, group 3 will receive cinnulin PF 500mg. Subjects will be instructed to take their study pills once a day for 90 days.After 90 days of treatment, each subject will again have hemoglobin A1C, lipid panel, height, weight, blood pressure and waist circumference measured. Analysis described above using intention-to-treat principles for any missing data will be used (we will use the carry-forward method to impute missing data). Subjects will bring in any remaining medication to determine adherence rates to the study protocol.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

* Patients 18 years or older.
* Diagnosed with type 2 diabetes mellitus within the past 30 days or who have been diagnosed and have not begun treatment.

Exclusion:

* Subjects who are <18 yrs of age.
* Pregnant or breastfeeding.
* Allergic to cinnamon.
* Allergic to metformin.
* Patients taking metformin are excluded from participating, unless they agree to wash out for two weeks prior to entering the study.
* Patients taking Cinnamon as a dietary supplement are excluded from participating, unless they agree to wash out for two weeks prior to entering the study.
* Patients taking any of the following:

  * Daily oral steroids
  * Warfarin
  * Hypoglycemic medication
  * Weight loss medication
  * Digoxin, lithium, phenytoin, & theophylline (due to narrow therapeutic indices)
* Serum creatinine >1.5 (this is standard of care that would be measured by PCM upon diagnosis of type 2 diabetes mellitus)
* Initial hemoglobin A1C >9.5(this is standard of care that would be measured by PCM upon diagnosis of type 2 diabetes mellitus).
* Clinical or laboratory evidence of liver disease.
* Clinical or laboratory evidence of Alcoholism.
* New York Heart Association (NYHA) Class III and IV congestive heart failure.

  * Class III: Cardiac disease resulting in marked limitation of physical activity - less than ordinary activity causes fatigue, palpitation, dyspnea, or angina. Comfortable at rest.
  * Class IV: Cardiac disease resulting in inability to carry on any physical activity without discomfort or symptoms. Symptoms may be present at rest. If any physical activity is undertaken, discomfort or symptoms are increased.
* Patients who are known to have or develop during the study any of the following upon review of their medical record:

  * Celiac disease
  * Insulinoma
  * Cushings Disease
  * Hyperthyroidism
  * Acromegaly
  * Phechromocytoma
  * Addison's Disease
  * Galactosemia
  * Glycogen storage disease
  * Hereditary fructose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, M.D., Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (1):
- Mike O'Callaghan Federal Hospital, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Cinnamon Bark | Cinnulin PF
Started | 7 | 8 | 10
Completed | 6 | 7 | 8
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Cinnamon Bark | Cinnulin PF | Total
Number analyzed (Participants) | 7 | 8 | 10 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 8 | 17
  >=65 years | 2 | 4 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 9
  Male | 4 | 4 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Decrease in HbA1c
Description: Subjects will have baseline blood levels to measure HbA1c. Subjects will then take either cinnamon bark powder, water-soluble cinnamon extract or metformin for 90 days then blood levels of HbA1c and lipid panel will be drawn again.
Time Frame: 90 days
Population: no data was analyzed as study was stopped early due to low recruitment
Arm/Group | Metformin | Cinnamon Bark | Cinnulin PF
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Decrease in LDL Cholesterol
Description: Subjects will have baseline blood levels to measure LDL Cholesterol. Subjects will then take either cinnamon bark powder, water-soluble cinnamon extract or metformin for 90 days then blood levels of HbA1c and lipid panel will be drawn again.
Time Frame: 90 days
Population: no data was analyzed as study was stopped early due to low recruitment
Arm/Group | Metformin | Cinnamon Bark | Cinnulin PF
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Metformin | Cinnamon Bark | Cinnulin PF
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes